CLINICAL TRIAL: NCT00763945
Title: Aachen Digital Myocardial Infarction Register
Brief Title: Infarction Register
Acronym: ADMIRE
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: PD Dr. med. Wolfgang Lepper, RWTH Aachen University, Medical Faculty
Other Study IDs: ADMIRE
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary Syndrome; STEMI; NSTEMI; Registry
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Data Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients representing to the hospital with acute coronary syndrome
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — The data of patients is collected from their hospital documentation The follow-up of all patients is done via phone calls in order to collect data about the outcome of each patient

SUMMARY:
The Aachener Digitale Myokardinfarkt Register (ADMIRE) is a prospektive registry study which was designed in order to obtain data of patients with acute coronary syndrome and herewith control and optimize guideline conform therapy of these patients.

DETAILED DESCRIPTION:
Aims of this registry stdy are

documentation of the characteristics of all patients representing to the RWTH Aachen University Hospital (UKA) with STEMI or NSTEMI documentation of the invasive and adjuvant medicinal therapy of STEMI and NSTEMI at UKA documentation of the in-hospital mortality documentation of the procedure-associated complications documentation of therapeutic principals for patients with STEMI or NSTEMI at UKA and investigation conformity of treatment with already established guidelines

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome

Exclusion Criteria:

* under age or not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the hospital with acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Verena Deserno, M.Sc., Study Director — Medical Faculty of the RWTH Aachen University; Rainer Hoffmann, MD, Ph.D., Principal Investigator — RWTH Aachen University Hospital
Locations (1):
- Department of Medicine, Division of Cardiology, Pulmonary Diseases and Vascular Medicine at the University Hospital, RWTH Aachen, Aachen, North Rhine-Westphalia, Germany